CLINICAL TRIAL: NCT03227601
Title: Effect of a Posture Adapter Use on Body Alignment in Standing Position on Children Between 12 and 24 Months Old With Zyka Virys Congenital Syndrome
Brief Title: Effect of a Posture Adapter for 12 to 24-month Children With Zyka Virus Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, Labibe Mara Pinel Frederico, master's student, Universidade Federal de Pernambuco
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1808
Record Dates: First submitted 2017-07-20; First posted 2017-07-24 (Actual); Last update posted 2017-07-24 (Actual); Status verified 2017-07

CONDITIONS: Zika Virus
MeSH Terms: conditions — Zika Virus Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: posture adapter — continued use of the device at home for 2 months after instructions of how to do it

SUMMARY:
Congenital Zika virus syndrome (SCZv) has been gaining attention in studies due to changes in the central nervous system and in the motor development of children. These changes resulted in an unexpected picture and without future predictability, with the appearance of several functional impairments and also on orthostatic posture. In this context, the protocol of orthostatism proposed here is a 10-week program of the use of a postural adjuster, the standing frame, made of its own with alternative material to the commercial models (cardboard). The use of low cost materials allows these devices to be made in the desired size without cost high, individually adapted, easy to be transported as it is light and can still be colored. It is an equipment that offers the opportunity to experience the orthostatic posture and mainly benefits children with little economic resources that enable the acquisition of traditional devices made of iron or wood and even imported equipment. The postural adjuster allows physical and sensorial opportunity, being an auxiliary resource in standing positioning, feasible for home use, besides being useful for performing functional activities. Thus, the objective will be to analyze the repercussions of the use of the standing frame on body alignment, muscle tone, gross motor function and gastrointestinal functions of children with SCZv. An uncontrolled intervention study will be conducted with children between 12 and 24 months of age, who will undergo an evaluation before use and after the use of the adjunct along with the proposed orthostatism protocol. The postural alignment will be evaluated through photogrammetry and the evaluation of muscle tone will be performed through the modified Tardieu scale. The Gross Motor Function Measure (GMFM) scale will be used to assess the gross motor function of the children involved in the study. Questionnaires will be applied for the collection of maternal socio-demographic data, the child's data, the type and time of therapy that the child already participates, and the gastrointestinal functions. Evaluations will occur in four moments: initial / before use, on the first day of placement in the adjuster, after the first month after use and after the second month of use. For statistical analysis, the Shapiro Wilk Test will be applied to evaluate the normality of the data, and the Friedman or ANOVA tests for repeated samples, to analyze intra-group time factor for the dependent variables of each individual.

ELIGIBILITY:
Inclusion Criteria:

* children between 12 and 24 months old;
* children with confirmed zika virus infection diagnosis;
* children with STORCH + for zika virus (blood test)

Exclusion Criteria:

* children with no medication for controlling zika virus infection symptoms;
* children with musculoskeletal disorders or limitation to standing position

Ages: 12 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2017-07-20 (Actual); Primary Completion 2017-10-19 (Estimated); Study Completion 2018-08-31 (Estimated)

PRIMARY OUTCOMES:
Body Alignment | two-month period
  Position or attitude of the body, the Arrangement of the parts of the body for a specific activity, or a Characteristic way of someone sustaining your body

SECONDARY OUTCOMES:
Motor function | two-month period
  Ability to carry out human development stages
Gastrointestinal function | two-month period
  intestinal motility
Muscular tonus | two-month period
  basal level of muscle contraction

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Federal de Pernambuco, Recife, Pernambuco, Brazil